CLINICAL TRIAL: NCT04379180
Title: Population Pharmacokinetics and Dosage Individualization of Bosentan, Sildenafil and Tadalafil in Persistent Pulmonary Hypertension of the Newborn
Brief Title: Population Pharmacokinetics and Dosage Individualization of Oral Pulmonary Vasodilators in PPHN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Collaborators: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: 2020_PPHN_001
Record Dates: First submitted 2020-04-26; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — Bosentan; Sildenafil Citrate; Tadalafil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment(bosentan, sildenafil and tadalafil)
  Interventions: Drug: Bosentan Tablets; Drug: Sildenafil Tablet; Drug: Tadalafil Tablets

INTERVENTIONS:
Drug: Bosentan Tablets — 2mg/kg, bid
Drug: Sildenafil Tablet — 1mg/kg, q6h/q8h
Drug: Tadalafil Tablets — 1mg/kg, qd

SUMMARY:
The use of bosentan, sildenafil and tadalafil in neonates with persistent pulmonary hypertension (PPHN) depends mostly on the empirical experience of pediatricians. Moreover, the recommended dose of those three drugs in treating PPHN remains controversial. Therefore, our aim is to study the pharmacokinetics and pharmacodynamics of bosentan, sildenafil and tadalafil in neonates of PPHN then dose a tailor-made therapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age: postnatal age ≤ 28 days;
* Patients have been diagnosed with PPHN;
* Bosentan, sildenafil and/or tadalafil used as part of regular treatment.
* Parental written consent

Exclusion Criteria:

* Expected survival time less than the treatment cycle;
* Major congenital malformations;
* Undergoing surgery within the first week of life;
* Receiving other systemic trial drug therapy;
* Other factors that the researcher considers unsuitable for inclusion.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates suffered from persistent pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-26 (Estimated); Primary Completion 2023-02-26 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Oxygenation index | The first 72 hours of the initial treatment
  Oxygenation index=(fraction of inspired oxygen*mean airway pressure)/the partial pressure of arterial oxygen
The change of hemodynamics | Through study completion, an average of 5 days
  * Pulmonary artery pressure (mmHg)
  * Alveolar-arterial gradient (mmHg)

SECONDARY OUTCOMES:
Duration of hospitalization | Within the first 28 days of patients' life
  Duration of initial therapy
Death | Within the first 28 days of patients' life
  Death in the first 28 days of life
Adverse events | Through study completion, an average of 5 days
  Drug-related adverse events and serious adverse events
Sequelae of PPHN | Through study completion and a 6-month visit
  Including cerebral palsy, hearing impairment, neurodevelopmental outcome etc
The need of extra support | Through study completion, an average of 5 days
  Besides the initial therapy (bosentan, sildenafil and/or tadalafil), other support such as inhaled nitric oxide (iNO), inotropic agents or Extracorporeal Membrane Oxygenation (ECMO)
Pulse oxygen saturation | The first 72 hours of the initial treatment
  Pulse oxygen saturation（%）

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided